CLINICAL TRIAL: NCT02226913
Title: Effect of Sodium Bicarbonate Buffered Lidocaine on the Success of Inferior Alveolar Nerve Block for Teeth With Symptomatic Irreversible Pulpitis: A Prospective, Randomized Double-blind Study
Brief Title: Effect of Sodium Bicarbonate Buffered Lidocaine on the Success of IAN Block of Teeth With Irreversible Pulpitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Masoud Saatchi (Other)
Responsible Party: Sponsor-Investigator, Masoud Saatchi, associate professor, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 193396
Record Dates: First submitted 2014-07-02; First posted 2014-08-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Local Anesthesia
Keywords: Buffered; inferior alveolar nerve block; irreversible pulpitis; local anesthesia; sodium bicarbonate
MeSH Terms: interventions — Lidocaine; Epinephrine; Septodont; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lidocaine & sodium bicarbonate (Experimental): 2% lidocaine with 1: 80,000 epinephrine buffered with 0.18 mL of 8.4% sodium bicarbonate
  Interventions: Drug: 2% lidocaine with 1:80,000 epinephrine; Drug: sodium bicarbonate
- lidocaine & placebo (Active Comparator): 2% lidocaine with 1:80,000 epinephrine with 0.18 mL of sterile distilled water
  Interventions: Drug: 2% lidocaine with 1:80,000 epinephrine; Drug: placebo

INTERVENTIONS:
Drug: 2% lidocaine with 1:80,000 epinephrine — 2% lidocaine with 1:80,000 epinephrine
  Other Names: Lignospan; Septodont, Saint Maur des Fosses, France
Drug: sodium bicarbonate — 8.4% sodium bicarbonate
  Other Names: Samen Laboratories (Mashhad, Iran)
  Arms: lidocaine & sodium bicarbonate
Drug: placebo — sterile distilled water (Samen Pharmaceutical Co, Iran)
  Other Names: sterile distilled water (Samen Pharmaceutical Co, Iran)
  Arms: lidocaine & placebo

SUMMARY:
Buffering of local anesthetics (alkalinization) has been suggested in achieving pain control. The purpose of this prospective, randomized, double-blind study was to evaluate the effect of adding 0.6 mL 8.4% sodium bicarbonate to 3.0 mL 2% lidocaine with 1: 80,000 epinephrine on the success rate of IAN block for endodontic treatment of mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Some studies have been shown buffering of local anesthetics reduce pain of injection, hasten the onset of anesthesia, and improved success rate of anesthesia. Others reported buffering of local anesthetics cannot reduce pain of injection, hasten the onset of anesthesia, and improve success rate of anesthesia. There are no studies evaluating a sodium bicarbonate-buffered lidocaine formulation for IAN block for teeth with irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* vital mandibular molar tooth
* diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* younger than 18 years old
* history of significant medical conditions
* allergies to local anesthetics or sulfites
* pregnancy
* taking any medications that might influence anesthetic assessment
* active sites of pathosis in area of injection
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of the success of IAN Block anesthesia with a buffered 2% lidocaine with 1:80,000 epinephrine solution for inferior alveolar nerve block | Baseline

SECONDARY OUTCOMES:
Heft-Parker visual analog scale recording of a non-buffered 2% lidocaine with 1:80,000 epinephrine solution for inferior alveolar nerve block | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Saatchi, DDS MSc, Study Chair — Isfahan University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No